CLINICAL TRIAL: NCT03128346
Title: Analgesic Effects of Transversus Thoracic Plane (TTP) Block in Cardiac Surgery - Pilot Study
Brief Title: Analgesic Effects of Transversus Thoracic Plane (TTP) Block in Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Satoru Fujii, Clinical fellow, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 109015
Record Dates: First submitted 2017-04-09; First posted 2017-04-25 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Postoperative Pain; Nerve Block; Cardiac Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone; Aspirin; Acetaminophen; Fentanyl

STUDY DESIGN:
Intervention Model Description: two groups: the nerve block group and the standard of care group
Who Masked: Participant
Masking Description: Participants will be blinded to the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The nerve block group (Experimental): TTP block under dynamic ultrasound guidance plus the standard care (hydromorphone, fentanyl, aspirin, acetaminophen)
  Interventions: Procedure: Transthoracic Transversus Plane Block; Drug: Hydromorphone Hydrochloride; Drug: Aspirin; Drug: Acetaminophen; Drug: Fentanyl
- The standard of care group (Active Comparator): Patients in the standard care group will receive pain medications, such as hydromorphone, fentanyl, aspirin and acetaminophen.
  Interventions: Drug: Hydromorphone Hydrochloride; Drug: Aspirin; Drug: Acetaminophen; Drug: Fentanyl

INTERVENTIONS:
Procedure: Transthoracic Transversus Plane Block — The investigator (RF or DV) will administer bilateral TTP block under dynamic ultrasound guidance with an echogenic needle using a total of 40mL of 0.5% ropivacaine (200mg), 20mL on each side. If the patient is less than 70kg, the total dose administered will be 40mL of 0.3% ropivacaine (150mg). The patient will not require sedation or analgesia for the performance of the block. The projected time for block completion is 20 minutes after appropriate patient positioning (supine) and exposure (upper chest). After block administration, the patient will be monitored for local anesthetics toxicity, hemodynamic instability, and allergic or unexpected adverse reactions for 20 minutes. Standard intensive care monitors are sufficient.
  Arms: The nerve block group
Drug: Hydromorphone Hydrochloride — IV, Hydromorphone
Drug: Aspirin — Oral Aspirin
Drug: Acetaminophen — Oral acetaminophen
  Other Names: tylenol
Drug: Fentanyl — IV, fentanyl

SUMMARY:
The TTP block is a novel regional anesthetic technique that shows promise in providing analgesia for anterior chest wall incisions and median sternotomy. The investigators hope to show that by providing the TTP block, there will be reduced early postoperative pain, reduced sedation and shallow breathing, reduced time on breathing machine, leading to an increase in patient comfort and satisfaction. The investigators also hope the decreased need for pain medication and reduced time on the breathing machine will translate into decreased nursing workload.

DETAILED DESCRIPTION:
In February 2015, Ueshima et al published an article regarding ultrasound guided transversus thoracic muscle plane (TTP) block for breast cancer resection. In this article, he showed that branches of the intercostal nerves (Th2-6) dominate the region of the internal mammary area. By administering local anesthetics between the internal intercostal and transversus thoracic muscle, analgesia in the anterior chest and sternum can be obtained. A cadaveric study shows injectate spread from the second to fifth intercostal spaces with a single 15mL injection between the third and fourth ribs next to the sternum. They further published a case series of two patients who successfully underwent median sternotomy for aortic valve replacement and thymoma resection using only the TTP block for analgesia. Fast- track cardiac surgery is now widely practiced, and evidence for its safety and efficacy has spurred its adoption. With the increased demand for health care resources including nursing manpower and ICU beds, postoperative patients are returning to the cardiac surgery intensive care unit (CSICU) on shorter acting anesthetic agents so that they can be awakened, following commands and spontaneously ventilating earlier. The TTP block fits in well with the fast- track paradigm. By providing adequate analgesia for median sternotomy, the TTP block may reduce narcotic requirements and consequent sedation and respiratory depression, hypercapnia and respiratory acidosis, prolonged mechanical ventilation and need for emergency advanced airway interventions.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgical procedures performed by a single conventional median sternotomy, and first case of the day patient because early postoperative pain scores are difficult to obtain overnight for patients admitted to the ICU in the evening.

Exclusion Criteria:

* patients undergoing non-median sternotomy access, surgeries involving saphenous vein or radial artery harvests, emergency cases, LVEF (Left ventricular efection fraction) <30%, ASAPS (American society of anesthesiologists physical status)=5, known local anesthetic allergy, allergy to any study medications, pre-existing major organ dysfunction including hepatic and renal failure, eGFR (estimated glomerular filtration rate) <60mL/min/1.73m2, coagulopathy, hematological disorders, infection at the site of injection, significant psychiatric illnesses (schizophrenia, bipolar, uncontrolled anxiety or depression), narcotic dependency (chronic opioid use of greater than 15mg oral morphine equivalents daily), peripheral neuropathy, pregnancy, patient refusal, lack of informed consent, moderate cognitive impairment, and language or reading barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Narcotic requirements equivalents | From the time of ICU admission up to 48 hours
  The amount of narcotics (hydromorphone or fentanyl) required will be assessed on patients' chart.

SECONDARY OUTCOMES:
Time to extubation | From the time of ICU admission up to 24 hours
  0 hour (the time of ICU admission) to extubation
Patient satisfaction satisfaction | From extubation up to 48 hours
  yes or no
Pain score equivalents | From the time of ICU admission up to 48 hours
  on a sclale of 0-10
Respiratory rate | After extubation up to 48 hours
  Every 2 hours after extubation
Oxygen saturation by pulse oximetry | After extubation up to 48 hours
  After extubation

OTHER OUTCOMES:
Recruitment rate | From the time of first recruitment up to one month
  Recruitment rate (Main outcome in the feasibility study, which will be conducted prior to the main study.)
Acceptability | From the time of ICU admission up to 48 hours
  Acceptability will be assessed using a likert scale questionnaire(Main outcome in the feasibility study, which will be conducted prior to the main study.)
Nausea/Vomiting | After extubation up to 48 hours
  Anti-emetics requirements

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ueshima H, Hara E, Marui T, Otake H. RETRACTED: The ultrasound-guided transversus thoracic muscle plane block is effective for the median sternotomy. J Clin Anesth. 2016 Mar;29:83. doi: 10.1016/j.jclinane.2015.10.014. Epub 2016 Feb 9. No abstract available. PMID 26897453
- [Result] Ueshima H, Otake H. Limitations of the Transversus Thoracic Muscle Plane Block. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):659-60. doi: 10.1097/AAP.0000000000000463. No abstract available. PMID 27547910 (Retraction: PMID 32571846 Reg Anesth Pain Med. 2020 Jun 22;:)
- [Result] Ueshima H, Kitamura A. Blocking of Multiple Anterior Branches of Intercostal Nerves (Th2-6) Using a Transversus Thoracic Muscle Plane Block. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):388. doi: 10.1097/AAP.0000000000000245. No abstract available. PMID 26079353
- [Result] Ueshima H, Otake H. Where is an appropriate injection point for an ultrasound-guided transversus thoracic muscle plane block? J Clin Anesth. 2016 Sep;33:190-1. doi: 10.1016/j.jclinane.2016.03.057. Epub 2016 May 1. No abstract available. PMID 27555162 (Retraction: PMID 35393189 J Clin Anesth. 2022 Aug;79:110733)
- [Derived] Fujii S, Roche M, Jones PM, Vissa D, Bainbridge D, Zhou JR. Transversus thoracis muscle plane block in cardiac surgery: a pilot feasibility study. Reg Anesth Pain Med. 2019 May;44(5):556-560. doi: 10.1136/rapm-2018-100178. Epub 2019 Mar 21. PMID 30902911